CLINICAL TRIAL: NCT03619902
Title: A Single Arm Multiple Dose Study to Assess the Efficacy and Safety of ANB019 in Subjects With Generalized Pustular Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in Adults With Generalized Pustular Psoriasis
Acronym: GPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANB019-002; 2017-004021-33 (EudraCT Number)
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-03

CONDITIONS: Generalized Pustular Psoriasis
Keywords: GPP
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imsidolimab (Experimental): Participants received imsidolimab 750 mg intravenously (IV) on Day 1 followed by administration of 3 doses of subcutaneous (SC) imsidolimab 100 mg on Days 29, 57, and 85.
  Interventions: Biological: Imsidolimab

INTERVENTIONS:
Biological: Imsidolimab — Humanized monoclonal antibody
  Other Names: ANB019

SUMMARY:
The main objectives of this study are to evaluate the efficacy, safety and tolerability of imsidolimab in adults with active GPP.

DETAILED DESCRIPTION:
Single arm, multiple-dose study evaluating the use of imsidolimab for the treatment of GPP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active GPP
* Japanese Dermatology Association (JDA) severity index total score of at least 6 and erythema with pustules accounting for at least 10% of body surface area or a moderate severity score on Generalized Pustular Psoriasis Physician's Global Assessment (GPPPGA)
* Must be candidates for systemic therapy or phototherapy

Exclusion Criteria:

* Erythrodermic, guttate psoriasis, drug induced GPP
* Any other ongoing inflammatory disease that interfere with the Investigator's ability to evaluate the subject's response to therapy
* History of recurrent or chronic infection
* ongoing use of psoriasis prohibited medication

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Site 102, Encino, California
  - Site 105, Largo, Florida
  - Site 104, Miami, Florida
  - Site 101, Indianapolis, Indiana
  - Site 100, Ann Arbor, Michigan
- Poland (4):
  - Site 303, Lodz
  - Site 302, Lodz
  - Site 304, Olsztyn
  - Site 301, Rzeszów
- Site 501, Seoul, South Korea
- United Kingdom (3):
  - Site 201, London
  - Site 203, Newcastle upon Tyne
  - Site 202, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers that enrolled subjects in the United Kingdom and Poland.
Pre-assignment Details: The study included a screening period of up to 42 days, a 12-week treatment period, and a 12-week safety follow-up period. A total of 12 subjects were screened, with 8 subjects being enrolled in the study.
Period: Overall Study
Arm/Group | Imsidolimab
Started | 8
Completed | 6
Not Completed | 2
Not completed — Termination of Study by Investigator | 1
Not completed — Use of Excluded/Prohibited Medication | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Imsidolimab: Participants received imsidolimab 750 mg intravenously on Day 1 followed by administration of 3 doses of subcutaneous imsidolimab 100 mg on Days 29, 57, and 85.
Arm/Group | Imsidolimab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 7
Region of Enrollment [Number; unit: participants]
  Poland | 5
  United Kingdom | 3
Modified Japanese Dermatological Association Severity Index (JDA-SI) Total Score [Mean (Standard Deviation); unit: score on a scale] — The JDA-SI includes assessment of skin lesions (area of erythema with pustules, area of erythema total, and area of edema) and fever, white blood cell count, C-reactive protein and serum albumin levels. The total score ranges from 0 to 17 (severe).
  score on a scale | 9.1 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response on the Clinical Global Impression (CGI) Scale
Description: Clinical response was defined as "Very much improved," "Much Improved," or "Minimally Improved" on the CGI scale according to the Modified Japanese Dermatological Association Severity Index (JDA-SI) total score.
  The JDA-SI includes assessment of skin lesions (area of erythema with pustules, area of erythema total, and area of edema) and fever, white blood cell count, C-reactive protein and serum albumin levels. The total score ranges from 0 to 17 (severe).
  CGI was assessed based on the JDA-SI according to the following:
  * Very Much Improved: Reduction in JDA-SI total score by 3 or > points;
  * Much improved: Reduction in JDA-SI total score by 1 or 2 points;
  * Minimally improved: No change in JDA-SI total score and area of erythema with pustules reduced by <20% or clinically meaningful improvement in at least 1 other component of the modified JDA-SI.
Time Frame: Week 4 and Week 16
Population: The full analysis set (FAS) included all enrolled participants. Participants with missing data were categorized as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imsidolimab
Number analyzed (Participants) | 8
percentage of participants
  Week 4 | 75.0 [34.91 to 96.81]
  Week 16 | 75.0 [34.91 to 96.81]

2. Primary Outcome: Percent Change From Baseline in Body Surface Area of Erythema With Pustules at Week 1, Week 4, and Week 16
Description: Excluding palms and soles from 0% to 100%. The palmar surface of one hand (using the subject's hand and including the fingers) represents 1% of his or her total BSA.
Time Frame: Baseline, Week 1, Week 4, and Week 16
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Imsidolimab
Number analyzed (Participants) | 8
percent change
  Week 1 | -59.63 (39.895)
  Week 4: number analyzed (Participants) | 6
  Week 4 | -94.17 (10.737)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -97.78 (5.443)

3. Secondary Outcome: Percent Change From Baseline in Modified Japanese Dermatological Association - Severity Index (mJDA-SI) Total Skin Lesions Score at Week 1, Week 4, and Week 16
Description: The area of erythema with pustules, area of total erythema and area of edema were assessed by the Investigator and scored from 0 to 3 on the following scale:
  * 0: 0% body surface area (BSA) affected;
  * 1: > 0%, < 10% BSA affected;
  * 2: ≥ 10%, < 50% BSA affected;
  * 3: ≥ 50% BSA affected.
  The JDA-SI Total Skin Lesions Score is the sum of the area of erythema with pustules score, area of total erythema score and area of edema score and ranges between 0 and 9 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 1, Week 4, and Week 16
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Imsidolimab
Number analyzed (Participants) | 8
percent change
  Week 1 | -25.74 (26.369)
  Week 4: number analyzed (Participants) | 6
  Week 4 | -55.65 (27.157)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -62.20 (29.757)

4. Secondary Outcome: Percentage of Participants Achieving a Generalized Pustular Psoriasis Physician's Global Assessment (GPPPGA) Score of 0 or 1 at Week 1, Week 4, and Week 16
Description: The GPPPGA scale was used to assess the impact and severity of GPP on the following scale:
  * 0: Clear (normal skin or post-inflammatory hyperpigmentation, no visible pustules, no scaling or crusting).
  * 1: Almost clear (faint, diffuse pink or slight red erythema, low density occasional small discrete pustules (noncoalescent), superficial focal scaling or crusting restricted to periphery of lesions).
  * 2: Mild (light red erythema, moderate density grouped discrete small pustules (noncoalescent), predominantly fine scaling or crusting).
  * 3: Moderate (bright red erythema, high density pustules with some coalescence, moderate scaling or crusting covering most or all lesions).
  * 4: Severe (deep fiery red erythema, very high density pustules with pustular lakes, severe scaling or crusting covering most or all lesions).
Time Frame: Week 1, Week 4, and Week 16
Population: Full Analysis Set participants with GPPPGA at Baseline and at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imsidolimab
Number analyzed (Participants) | 5
percentage of participants
  Week 1 | 0.0 [0.00 to 52.18]
  Week 4: number analyzed (Participants) | 4
  Week 4 | 50.0 [6.76 to 93.24]
  Week 16: number analyzed (Participants) | 4
  Week 16 | 75.0 [19.41 to 99.37]

5. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 1, Week 4, and Week 16
Description: The DLQI is a 10-item questionnaire that asks participants to evaluate the degree that their skin problem has affected their quality of life in the last week in the following 6 aspects: symptoms and feelings, daily activities, leisure, work or school activities, personal relationships and treatment related feelings. Participants answer the 10 questions on a scale from 0 (not at all) to 3 (very much). The DLQI is calculated by summing the scores of the 10 questions, resulting in a maximum of 30 and a minimum of 0 with higher scores indicating more impaired quality of life. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 1, Week 4, and Week 16
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imsidolimab
Number analyzed (Participants) | 8
score on a scale
  Week 1 | -0.9 (0.356)
  Week 4: number analyzed (Participants) | 6
  Week 4 | -6.0 (9.08)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -10.7 (9.16)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to end of follow-up period; 24 weeks.
Arm/Group | Imsidolimab
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imsidolimab (N=8)
COVID-19 (Infections and infestations) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imsidolimab (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (3)
Blood folate decreased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Myxomatous mitral valve degeneration (Cardiac disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish trial results until after the first multi-center publication unless such publication is not published within a period that is at least 18 months but less than or equal to 24 months after trial completion. In addition, the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03619902/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT03619902/SAP_001.pdf